CLINICAL TRIAL: NCT04630093
Title: Clinical Implementation Pilot of Preemptive Pharmacogenetic Testing in Medically Underserved Patient Populations
Brief Title: Pilot of Preemptive Pharmacogenetics in Medically Underserved Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202002594-N; UL1TR001427 (NIH)
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pharmacogenetic Testing
Keywords: Pharmacogenetics; Medically underserved; Implementation; Effectiveness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Panel-based pharmacogenetic genotyping (Experimental): All patients will receive clinical preemptive pharmacogenetic testing. Genotype results and consult notes will returned in the EHR pre-emptively. Data on implementation success metrics and PROs via patient report and TSQM measures will be collected. In addition, data on effectiveness outcomes and socioeconomic measures will be collected via the EHR and patient report, respectively.
  Interventions: Diagnostic Test: Panel-based pharmacogenetic genotyping

INTERVENTIONS:
Diagnostic Test: Panel-based pharmacogenetic genotyping — A DNA sample by saliva (via mouthwash swish and expectorate collection) or buccal cell (via buccal brush) will be obtained for pharmacogenetic testing and questionnaires will be administered at baseline and then again at 3 months and 6 months after receiving PGx results.

SUMMARY:
This is a pragmatic clinical trial of 100 patients who self-identify as black or Latino. Patients with active prescriptions for at least 3 medications and a medication change within the past 6-months will be recruited from the University of Florida (UF) Health primary care clinics for panel-based pharmacogenetic testing. Participants will be followed for 6 months and will undergo assessments with the Treatment Satisfaction Questionnaire for Medication (TSQM) three times (baseline visit, 3-month visit, and 6-month visit post pharmacogenetic testing). In addition, data on effectiveness outcomes and socioeconomic measures will be collected via the electronic health record (EHR) and patient report. Participation is expected to last approximately 6 months and the study will be open for approximately 12-14 months.

DETAILED DESCRIPTION:
Little information exists regarding clinical implementation of pharmacogenetics in medically underserved patient populations. Preliminary data indicate that underserved patients are prescribed a higher rate of drugs associated with pharmacogenetic guidelines (pharmacogenetic drugs). Thus, an important knowledge gap exists regarding the use of pharmacogenetic in a patient population that may be the most likely to clinically benefit. The objective of this study is to develop key feasibility data to equitably advance preemptive pharmacogenetic testing within UF Health, and to generate important preliminary data to support future larger studies. This objective will be accomplished by pursuing three specific aims: (1) assess the feasibility of preemptive pharmacogenetic clinical implementation in primary care clinics predominantly serving medically underserved patients; (2) understand perspectives about preemptive pharmacogenetic among key stakeholders in the primary care clinics predominantly serving medically underserved patients; and (3) identify specific socioeconomic characteristics most strongly associated pharmacogenetic drug prescription rate.

One hundred patients who self-identify as black or Latino with active prescriptions for at least 3 medications, one of which can be informed by panel-based pharmacogenetic testing, and a medication change within the past 6-months will be recruited from UF Health primary care clinics for panel-based pharmacogenetic testing. Participants will be followed for 6 months and will undergo assessments with the Treatment Satisfaction Questionnaire for Medication (TSQM) three times (at baseline and then again during the 3and 6-month follow-up post pharmacogenetic testing). In addition, data on effectiveness outcomes and socioeconomic measures will be collected via the EHR and patient report. Records for patients receiving care at UF Health primary care clinics will be screened based on inclusion/exclusion criteria for participation in the study. Those that meet criteria will be offered participation. Participation is expected to last approximately 6 months and the study will be open for approximately 12-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) with active prescriptions for at least 3 medications documented within the EHR.
* At least 1 drug/drug class that could be informed by the pharmacogenetics test panel available at the UF.
* A medication change within the past 6 months (associated with a healthcare provider encounter).
* Self-identify as black or Latino.

Exclusion Criteria:

* Patients with any history of pharmacogenetic testing within the EHR.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Duarte, PharmD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panel-based Pharmacogenetic Genotyping
Started | 100
Completed | 99
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Panel-based Pharmacogenetic Genotyping
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 86
  White | 10
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 99
Reported annual household income [Count of Participants; unit: Participants]
  Less than $25,000 | 28
  $25,001-$50,000 | 20
  $50,001-$75,000 | 3
  $75,001-$100,000 | 3
  Greater than $100,000 | 1
  Unknown | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Patient Treatment Satisfaction Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The primary feasibility outcome will be change in patient treatment satisfaction between baseline and 6 months after pharmacogenetic testing. This patient reported outcome will be measured via the TSQM. The TSQM is a validated tool that assesses three medication-related domains (effectiveness, side effects, and convenience) to synthesize a global satisfaction score. TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction for that each domain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panel-based Pharmacogenetic Genotyping
Number analyzed (Participants) | 99
score on a scale
  Baseline | 59.9 (16.9)
  6 months | 64.4 (13.6)
Statistical Analysis 1: Comparison: Panel-based Pharmacogenetic Genotyping; Baseline vs. 6 months after receiving panel-based pharmacogenetic testing; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Patient Treatment Effectiveness Satisfaction Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: Change in patient treatment effectiveness satisfaction between baseline and 6 months after pharmacogenetic testing. This patient reported outcome will be measured via the TSQM. The TSQM is a validated tool that assesses three medication-related domains (effectiveness, side effects, and convenience) and a global satisfaction score. TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction for that each domain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panel-based Pharmacogenetic Genotyping
Number analyzed (Participants) | 99
score on a scale
  baseline | 59.6 (14.4)
  6 months | 63.3 (11.7)

3. Secondary Outcome: Change in Patient Treatment Side Effect Satisfaction Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: Change in patient treatment side effect satisfaction between baseline and 6 months after pharmacogenetic testing. This patient reported outcome will be measured via the TSQM. The TSQM is a validated tool that assesses three medication-related domains (effectiveness, side effects, and convenience) and a global satisfaction score. TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction for that each domain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panel-based Pharmacogenetic Genotyping
Number analyzed (Participants) | 99
score on a scale
  baseline | 84.2 (24.0)
  6 months | 85.5 (24.0)

4. Secondary Outcome: Change in Patient Treatment Convenience Satisfaction Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: Change in patient treatment convenience satisfaction between baseline and 6 months after pharmacogenetic testing. This patient reported outcome will be measured via the TSQM. The TSQM is a validated tool that assesses three medication-related domains (effectiveness, side effects, and convenience) and a global satisfaction score. TSQM domain scores range from 0 to 100 with higher scores representing higher satisfaction for that each domain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panel-based Pharmacogenetic Genotyping
Number analyzed (Participants) | 99
score on a scale
  baseline | 67.7 (13.2)
  6 months | 70.1 (11.7)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Panel-based Pharmacogenetic Genotyping
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04630093/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04630093/ICF_001.pdf